CLINICAL TRIAL: NCT01957878
Title: A Double-blind, Randomised, Placebo-controlled, Phase II Study to Evaluate ProCervix Efficacy to Clear HPV 16 and HPV 18 Infection in Women With Normal Cytology or ASCUS/LSIL
Brief Title: Phase II Study of HPV Therapeutic Vaccine in HPV Infected Women With Normal Cytology or ASCUS/LSIL
Acronym: RHEIA-VAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genticel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PC10VAC02
Record Dates: First submitted 2013-10-04; First posted 2013-10-08 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-12

CONDITIONS: Genital Infection Viral; HUMAN PAPILLOMA VIRUS

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HPV therapeutic vaccine (Experimental): ProCervix consists of two recombinant adenylate cyclase (CyaA) proteins, CyaA-HPV 16E7 (C16-1) and CyaA-HPV 18E7 (C18-1) in a 50/50 ratio (C16C18-2 Ag mixture). ProCervix is adjuvanted by Aldara™, a cream containing 5% of imiquimod
  Interventions: Biological: ProCervix
- Placebo matching ProCervix (Placebo Comparator): Placebo matching ProCervix and adjuvanted by Aldara™, a cream containing 5% of imiquimod
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ProCervix — ProCervix consists of two recombinant adenylate cyclase (CyaA) proteins, CyaA-HPV 16E7 (C16-1) and CyaA-HPV 18E7 (C18-1) in a 50/50 ratio (C16C18-2 Ag mixture). ProCervix is adjuvanted by Aldara™, a cream containing 5% of imiquimod
  Arms: HPV therapeutic vaccine
Biological: Placebo — Placebo matching ProCervix and adjuvanted by Aldara™, a cream containing 5% of imiquimod
  Arms: Placebo matching ProCervix

SUMMARY:
Human Papillomavirus (HPV) 16 and HPV 18 (the two virus genotypes targeted by the ProCervix vaccine) are the most common HPV genotypes associated with at least 70% of squamous cell carcinomas and 82% of adenocarcinomas of the cervix The strategy of therapeutic vaccination with ProCervix is to activate and enhance the patient's cellular immune response to HPV . The therapeutic vaccine will be used for women infected by HPV 16, HPV 18, or both. The vaccine targets these HPV infected women with normal or mild cervical cellular dyskaryosis as detectable infections with oncogenic potential.

This will be a double-blind, randomised, placebo-controlled, parallel group study assessing the efficacy of ProCervix or placebo (concomitantly administered with imiquimod cream).

ProCervix will be delivered with a topical agent, imiquimod, applied to the injection sites as a vaccine adjuvant.

The population proposed for this study represents an otherwise healthy female population who are infected with HPV 16 and/or HPV 18. The safety and tolerability of this therapeutic vaccine has been shown in the ongoing Phase I study, and the proposed population may in theory derive benefit from this vaccine.

ELIGIBILITY:
Inclusion Criteria:

* A subject will be eligible for inclusion in this study if the following criteria apply:

  1. Subject is female between the ages of 25 and 50 years (inclusive).
  2. Subject is pre-menopausal .
  3. Subject must have cervical HPV 16 and/or 18 infection confirmed by RT-PCR
  4. Subject has a cervical cytological evaluation with a normal, ASCUS or LSIL result at baseline.
  5. Subject has employed highly effective contraception the month prior to the first vaccination and will agree to employ highly effective contraception for at least 12 months after the first vaccination. .
  6. Subject is in general good health based on medical history and physical examination.
  7. Subject is able to communicate effectively with study personnel and is considered reliable, willing, and cooperative in terms of compliance with the protocol requirements.
  8. Subject voluntarily gives written informed consent to participate in the study.

Exclusion Criteria:

1. Subject has a current acute or chronic disease, other than infection with HPV, which would be expected to interfere with the planned evaluations of response
2. Subject has vaginal atrophy with or without topical hormonal therapies or systemic selective estrogen receptor modulators (SERMs).
3. Subject has prior exposure to HPV prophylactic vaccine or subject has participated in the past in another vaccination clinical trial related to infection with HPV
4. Current high grade lesions or history of untreated high grade cervical lesion (either CIN2 or CIN3).
5. Subject has current or a history of cancer of the cervix.
6. Subject has clinically significant (CS) gynaecological abnormalities that could interfere with study evaluation, in the judgment of the Investigator (e.g. prolapse, myoma, fibroid, hysterectomy).
7. Subject has a laboratory abnormality Grade ≥ 2, as defined using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventative Vaccine Clinical Trials,
8. Subject has received any live viral vaccine within 3 months or any other non live vaccine within 2 weeks of first study product administration.
9. Subject has primary or secondary systemic immunosuppression
10. Subject has a history of severe allergy (requiring hospital care) or history of severe asthma
11. Subject has a history of malignant cancer, except the following adequately treated cancers: basal cell carcinoma, or dermatological squamous cell carcinoma.
12. Subject was administered with another investigational drug or vaccine within 30 days prior to the screening visit or is participating in any other study.
13. Subject has a known hypersensitivity to imiquimod.
14. Subject has a history of severe reaction to any drug or vaccination.
15. Subject has a medical condition with clinical and/or biological consequences judged by the Investigator incompatible with vaccination(s).
16. Subject has positive results for human immunodeficiency virus (HIV), hepatitis B virus (HBV) surface antigen (HBsAg), or hepatitis C virus (HCV).
17. Subject has a symptomatic vaginal or genital infection
18. Subject has a history of or currently active genital herpes disease.
19. Subject is pregnant or is breastfeeding.
20. Subject has a positive serum human chorionic gonadotrophin (HCG) result at enrolment.

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 239 (Actual)
Dates: Start 2013-12; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Clearance of HPV 16 and HPV 18 infection at Month 12 using a type specific, sensitive and quantitative HPV PCR assay. | month 12

SECONDARY OUTCOMES:
Clearance of HPV 16 and HPV 18 infection. | Month 6, 15, 18, 24

CONTACTS AND LOCATIONS:
Locations (40):
- Belgium (4):
  - Regionaal Ziekenhuis Heilig Hart Tienen Hospital, Tienen, Vlaams Brabant
  - Centre for the Evaluation of Vaccination Vaccine & Infectious Disease Institute (VAXINFECTIO) Faculty of Medicine University of Antwerp Belgium, Antwerp
  - Grand Hôpital de Charleroi Site Notre-Dame, Charleroi
  - University Hospitals Leuven, Leuven
- Finland (3):
  - Helsinki University Central Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - Tampereen yliopistollinen sairaala Hospital, Tampere
- France (10):
  - CHU Amiens Hopital Sud, Amiens
  - Hôpital Saint Jacques, Besançon
  - GORH, CHU Estaing, Clermont-Ferrand
  - CHU Dijon, Dijon
  - Hôpital Jeanne de Flandre CHU de Lille, Lille
  - CHU de Nîmes - Hopital Universitaire Caremeau, Nîmes
  - Centre d'Investigation Clinique de Vaccinologie Cochin Pasteur (CIC BT505), Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Reims Institut Alix de Champagne, Reims
  - Hôpital de Hautepierre, Strasbourg
- Germany (6):
  - Charité - Universitätsmedizin Berlin Hospital, Berlin
  - Universitätsklinikum Erlangen Hospital, Erlangen
  - Elisabeth Krankenhaus Essen GmbH - Clinic/Outpatient Facility, Essen
  - Klinikum der Friedrich Schiller Universität Jena Hospital, Jena
  - LMU Klinikum der Universität- Hospital, München
  - Klinikum Wolfsburg Hospital, Wolfsburg
- Netherlands (2):
  - Center Gynaecological Oncology Amsterdam AMC, NKI-AVL, VUmc, Amsterdam
  - St. Antonius Ziekenhuis Hospital, Nieuwegein
- Spain (10):
  - Hospital Clinic Dept of Obstetrics and Gynecology C/ Villarroel Unidad de Ginecología Oncológica, Instituto Clínico de Ginecología y Obstetricia y Neonatología (ICGON), Hospital Clínic, Instituto de Investigaciones Biomédi, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall D Hebron, Barcelona
  - Institut Catala d'Oncologia L'Hopitalet de Llobregat, Barcelona
  - Clinica Ginecologica Ceoga, Clinic/Outpatient Facility, Lugo
  - Hospital Clínico San Carlos, Madrid
  - Hospital La Paz de Madrid, Madrid
  - Hospital Universitario "12 de Octubre", Madrid
  - Hospital Regional Universitario Carlos Haya - Hospital Materno Infantil, Málaga
  - Hospital Sagrado Corazón de Sevilla, Seville
- United Kingdom (5):
  - Dumfries and Galloway Royal Infirmary Hospital, Dumfries
  - Liverpool - GUM - Liverpool Centre for Sexual Health, Liverpool
  - St Mary's Hospital, London
  - Academic O&G University of Manchester Research - St Mary's Hospital, Manchester
  - The Centre for Immunology and Infection Hull York Medical School University of York, York